CLINICAL TRIAL: NCT06905834
Title: A Phase IIB Clinical Trial to Evaluate the Efficacy and Safety of Allogenic Mesenchymal Stem Cell (MSC) Injection Therapy for Refractory Graft-versus-Host Disease (GVHD) Unresponsive to Conventional Treatments
Brief Title: Evaluation of Allogenic Mesenchymal Stem Cell (MSC) Injection Therapy for Refractory Graft-versus-Host Disease (GVHD) Unresponsive to Conventional Treatments
Acronym: TER-EYE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto de Investigación Biomédica de Salamanca (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network); Instituto Universitario de Oftalmobiología Aplicada (Institute of Applied Ophthalmobiology) - IOBA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TERAV_24-01_EICRxEYE; 2024-519772-10-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-10; First posted 2025-04-01 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Dry Eye Disease (DED); Graft-Versus-Host Disease(GVHD)
Keywords: dry eye disease; Graft-versus-Host Disease; mesenchymal stem cells
MeSH Terms: conditions — Dry Eye Syndromes; Graft vs Host Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 6.25 million ASCs / 2,5ml of Ringer Lactato + 1% of HSA. (Experimental): 6.25 million mesenchymal cells will be injected subconjunctivally into each subject in the group. These cells will be in a 2.5 mL suspension of Lactated Ringer's solution, to which 1% HSA will have been added beforehand.
  Interventions: Drug: Subconjuntival injection of expanded allogenic adult adipose tissue-derived mesenchymal stem cells (ASC
- 12.5 million ASCs / 2,5 ml of Ringer Lactato + 1% of HSA. (Experimental): 12.5 million mesenchymal cells will be injected subconjunctivally into each subject in the group. These cells will be in a 2.5 mL suspension of Lactated Ringer's solution, to which 1% HSA will have been added beforehand.
  Interventions: Drug: Subconjuntival injection of expanded allogenic adult adipose tissue-derived mesenchymal stem cells (ASC

INTERVENTIONS:
Drug: Subconjuntival injection of expanded allogenic adult adipose tissue-derived mesenchymal stem cells (ASC — Subconjunctival injection is a widely used technique in ophthalmology due to its effectiveness, minimal invasiveness, and ease of administration. In a subconjunctival injection the cells adult adipose tissue-derived mesenchimal cells are delivered into the subconjunctival space, the area between the conjunctiva and sclera.

SUMMARY:
This Phase IIB, multicenter, double-blind, randomized, and uncontrolled clinical trial aims to assess the efficacy and safety of subconjunctival injection of Mesenchymal Stem Cells (MSCs) in patients with Graft-versus-Host Disease (GVHD) and severe ocular involvement (DYD-dry eye disease). The primary objective is to evaluate the clinically and statistically significant improvement in the signs and symptoms associated with the disease.

Secondary objectives include:

* Analyzing adverse events related to the subconjunctival injection of MSCs to confirm the safety of this treatment in patients with GVHD ocular involvement.
* Identifying new biomarkers that can be used to objectively assess the progression of patients with GVHD and severe ocular involvement.
* Studying the relationship between the expression of ocular surface-specific markers by MSCs and their clinical efficacy, as well as the variation in the expression of these markers in relation to cell preservation methods.

Assessing the quality of life of patients treated with two doses of MSCs using the NEI VFQ-25 (National Eye Institute Visual Function Questionnaire).

- Evaluating whether the cell dose impacts clinical improvement.

The trial includes 30 patients, divided into two groups of 15, and focuses on the assessment of dry eye disease, with the treatment based on MSC administration to improve clinical outcomes and quality of life for the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age who understand and sign the informed consent form.
* Diagnosis of severe GVHD (graft versus host disease) according to NIH criteria (revised by Lee SJ in 2017) with ocular involvement in the form of severe SOD (severe ocular disease) in both eyes for more than 3 months, objectively defined as superficial punctate keratitis >2 on the Oxford scale (range 0-5) and/or the presence of epithelial defect, and subjectively as severe symptoms, >33 points on the OSDI questionnaire (0-100).
* Patients must have previously been treated for at least three months with blood derivatives and/or insulin eye drops and topical cyclosporine or tacrolimus (unless any of these treatments were not tolerated and had to be discontinued).
* Patients must be using ocular lubricants at least 4 times a day and, despite this, still meet the criteria for severe SOD as outlined in point 2.
* Patients on low doses of topical corticosteroids for maintenance should have a stable dose for at least one month prior to inclusion.
* The dose and frequency of all topical medications the patient begins the trial with must remain unchanged throughout the duration of the trial, unless otherwise judged by the investigator.
* The chronic GVHD systemic treatment should be stable regarding the use of systemic immunosuppressors for at least one month prior to patient inclusion or before starting treatment.
* Negative result in the urine pregnancy test at the baseline visit for women of childbearing age. Subjects must be advised to use contraceptive methods during their participation in the clinical trial and undergo a new pregnancy test at the treatment visit if more than 28 days have passed since the baseline visit.

Exclusion Criteria:

* Uncontrolled systemic disease or any condition that, in the medical judgment, could put the patient at risk or affect the interpretation of the results.
* Uncontrolled systemic GVHD.
* Active ocular infection.
* Ocular surgery within the last 3 months.
* Initiation of topical therapies for SOD indicated in the inclusion criteria less than 3 months prior to inclusion.
* Start of topical corticosteroid use within 4 weeks prior to inclusion.
* Cognitive impairments that could interfere with study compliance.
* Pregnant women or women during the lactation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Change in the integrity of the ocular surface | six and twelve months from start of treatment
  Significant improvement in the integrity of the ocular surface, measured by corneal staining with fluorescein. A clinically significant improvement is defined as an improvement in Superficial Punctate Keratitis (SPK) of at least one unit compared to baseline, according to the Oxford scale (range 0-5). If an epithelial defect is present, a reduction of at least ¾ of its initial size is required. The Oxford scale is a grading system used to assess ocular surface damage based on corneal and conjunctival staining with fluorescein or lissamine green dyes. It is commonly used to evaluate conditions like dry eye disease and superficial punctate keratitis (SPK). The scale ranges from 0 to 5, where 0 represents no staining (healthy eye) and 5 indicates severe staining and damage.
Change in tear production | six and twelve months from start of treatment
  Significant increase in tear production, evaluated using the Schirmer test with topical anesthesia, by at least 2 mm. The Schirmer test is a diagnostic test used to measure tear production and assess dry eye syndrome. It evaluates whether the eyes produce enough tears to keep them properly lubricated. Results are as follows:
  Normal: ≥10 mm of wetting after 5 minutes Mild to moderate dry eye: 5-10 mm Severe dry eye: ≤5 mm
Change in the degree of conjunctival hyperemia | six and twelve months from start of treatment
  Significant reduction in the degree of conjunctival hyperemia by at least one point (Efron scale, 0-4). The Efron Scale is a clinical grading scale used by eye care professionals to assess the severity of contact lens complications and ocular surface conditions. It provides a standardized way to evaluate changes in the cornea and conjunctiva. The scale ranges from 0 to 4, where:
  Grade 0 = Normal (No signs of damage) Grade 1 = Trace (Mild changes, barely noticeable) Grade 2 = Mild (Early signs of irritation or damage) Grade 3 = Moderate (Significant changes, requires attention) Grade 4 = Severe (Serious complications, may need treatment)
Change in the parameters related to the Meibomian glands | six and twelve months from start of treatment
  Significant improvement, by at least one point, in parameters related to the Meibomian glands. The Meibomian glands are specialized sebaceous glands located in the upper and lower eyelids, near the edges of the eyelids. They are crucial for maintaining the health of the ocular surface. When the Meibomian glands become blocked or inflamed, it leads to Meibomian Gland Dysfunction (MGD). This condition can result in Dry eye disease. It is measured using Efron scale. The scale ranges from 0 to 4, where:
  Grade 0 = Normal (No signs of damage) Grade 1 = Trace (Mild changes, barely noticeable) Grade 2 = Mild (Early signs of irritation or damage) Grade 3 = Moderate (Significant changes, requires attention) Grade 4 = Severe (Serious complications, may need treatment)
Change in any of the findings in the central cornea | six and twelve months from start of treatment
  Significant improvement in any of the findings in the central cornea, evaluated through in vivo confocal microscopy:
  1. Improvement of at least one grade (three grades: corneal, mixed, conjunctival) in the epithelial phenotype.
  2. Significant reduction in the density of dendritic cells in the corneal stroma.
  3. Improvement in the characteristics of the sub-basal corneal nerve plexus (number of nerves, density, length, tortuosity, and nerve branching).
  All parameters are evaluated at the same time using the same samples, which will be analyzed by confocal microscopy.
Severity of eye disease measured by WFPRS (Wong-Baker Faces Pain Rating Scale) | six and twelve months from start of treatment
  The Wong-Baker Faces Pain Rating Scale (WFPRS) is a visual pain assessment tool that uses facial expressions to help individuals describe their pain intensity. The scale consists of six faces, ranging from a happy face (no pain) to a crying face (worst pain possible). Each face corresponds to a numerical value from 0 to 10:
  0-No Pain: The patient experiences no discomfort or pain and feels completely normal.
  2-Mild Pain: Slight discomfort is present but does not interfere with daily activities. No treatment necessary.
  4-Moderate Pain: Noticeable pain or discomfort, which may cause mild difficulty in performing certain tasks but is still manageable.
  6-Moderate to Severe Pain: Pain is more persistent and begins to interfere with concentration and daily functions. Medical attention may be needed.
  8-Severe Pain: Significant pain that affects daily activities and requires immediate medical attention.
  10-Worst Pain Possible: Extreme, unbearable pain that severily limits function.
Severity of eye disease measured by Numerical Rating Scale (NRS) | six and twelve months from start of treatment
  The Numerical Rating Scale (NRS) is a simple and widely used tool for assessing pain or symptom severity in patients. It typically asks individuals to rate their symptoms on a scale from 0 to 10, where:
  0 = No symptoms (or no pain) 10 = Worst possible symptoms (or unbearable pain)
  In dry eye assessments, the NRS is often used to rate:
  Eye dryness (0 = no dryness, 10 = extreme dryness) Eye discomfort (0 = no discomfort, 10 = severe discomfort)
  It helps track symptom progression and evaluate treatment effectiveness over time.
Severity of eye disease measured by Modified Symptom Assessment in Dry Eye Questionnaire (mSIDEQ) | six and twelve months from start of treatment
  The Modified Symptom Assessment in Dry Eye Questionnaire (mSIDEQ) is a patient-reported questionnaire used to assess the severity and impact of dry eye disease (DED) symptoms. It is an improved version of the original Symptom Assessment in Dry Eye Questionnaire (SIDEQ) and is designed to be more concise and clinically relevant. Patients rate their symptoms on a numerical scale (e.g., 0-4 or 0-5, depending on the version).
  The total score reflects the overall burden of dry eye symptoms-higher scores indicate worse symptoms.
Severity of eye disease measured by Ocular Surface Disease Index (OSDI) | six and twelve months from start of treatment
  The Ocular Surface Disease Index (OSDI) is a questionnaire used to assess the severity of dry eye disease (DED) and other ocular surface disorders. It evaluates the frequency of dry eye symptoms, their impact on daily activities, and environmental triggers that might worsen the condition. The OSDI consists of 12 questions divided into three categories:
  * Ocular Symptoms (e.g., dry eye discomfort, grittiness, pain)
  * Visual Function (e.g., difficulty reading, driving, using a computer)
  * Environmental Triggers (e.g., sensitivity to wind or air conditioning)
  Each question is scored from 0 to 4 (0 = no problems, 4 = severe problems). the results are analised as follows:
  0-12 → Normal 13-22 → Mild dry eye 23-32 → Moderate dry eye 33-100 → Severe dry eye
Severity of eye disease measured by CDES-Q (Contact Lens Dry Eye Symptom Questionnaire) | six and twelve months from start of treatment
  The Contact Lens Dry Eye Symptom Questionnaire (CDES-Q) is a patient-reported questionnaire designed to assess dry eye symptoms in contact lens wearers. It helps evaluate symptom severity, frequency, and impact on daily activities to better understand and manage contact lens-related dry eye (CLDE). Patients typically rate the frequency and severity of symptoms like:
  * Dryness or discomfort while wearing lenses
  * Burning or stinging sensations
  * Foreign body sensation (feeling like something is in the eye)
  * Blurred vision or fluctuating clarity
  * Lens awareness or intolerance over time Higher scores indicate more severe dry eye symptoms related to contact lens wear.

SECONDARY OUTCOMES:
Rate of adverse events related to the administration of subconjunctival ASC injection. | Through study completion, an average of 1 year
  The investigator will record in the eCRF and communicate to the sponsor or to the person assuming the tasks delegated by the sponsor, the adverse events (AEs) that are considered of special interest occurring during the study as soon as possible, and no later than 15 days after becoming aware of them.
  The AEs considered of special interest are:
  Immunogenicity reactions and their consequences. Adverse events possibly due to unexpected reactions such as hypersensitivity, immunological, toxic reactions, and migration of cells from the application site.
  Adverse events related to product failure that may be associated with the production process or with the quality of the investigational product.
Analysis of ocular marker expression in the administered ASCs | When vials are thawed before treating the first patients with 6.25 mill and 12.5 mill ASC, 1 year afterwards and two years afterwards or altertatively, when vials are thawed to treat the last patient with 6.25 and 12.5 mill ASC.
  The expression of the markers cytokeratin K3 and K12, specific to differentiated corneal epithelium, and the markers K15, nuclear transcription factor p63alpha (p63alpha), and ABCG2 transporter protein, specific to limbal corneal epithelium markers, will be analyzed using an immunodetection technique (immunofluorescence). It will also be analyzed how the freezing process of ASCs may affect these markers and, if possible, establish a correlation between the expression of these markers in the applied cells and the clinical outcomes.
Analysis of the presence and concentration of inflammation-related molecules in tear and serum samples | Visit 2 (day 14 ± 7 after screening), 6 months, 12 months and when applicable, at premature withdrawal.
  The presence and concentration of 48 inflammation-related molecules in tear and serum samples will be studied using the "Human Cytokine/Chemokine/Growth Factor Panel Cat. No. HCYTA-60KPXBK48" kit and XMAP™ technology (Luminex Corporation, Austin, TX, USA). All molecules are analyzed simultaneously, and their concentrations are measured in the same units, allowing for a combined analysis.
Search for new biomarkers that can be used to objectively evaluate the progression of patients affected by EICRc with ocular involvement. | Visit 2 (day 14 ± 7 after screening), 6 months, 12 months and when applicable, at premature withdrawal.
  The search for biomarkers aims at the development of predictive models that help improve the diagnosis of EICRc and the prognosis of these patients based on the expression of certain genes.

CONTACTS AND LOCATIONS:
Overall Officials: Fermín Sánchez-Guijo Martín MD, PhD, Medical Degree in Haematology, Study Director — Centro Asistencial Universitario de Salamanca (CAUSA); Lourdes Vázquez López MD, PhD, Medical Degree in Haematology, Principal Investigator — Centro Asistencial Universitario de Salamanca (CAUSA); Mi Kwon MD, PhD, Medical Degree in Haematology, Principal Investigator — Hospital General Universitario Gregorio Marañón (HGUGM)

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest (non-commercial interest) in advanced therapy in eye pathology, as dry eye. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Access Criteria: Any qualified researcher with academic interest migh ask acces to IPD after previous approval of the request by the project manager.